CLINICAL TRIAL: NCT06279221
Title: Litfulo® Capsules Special Investigation
Brief Title: Litfulo Capsules Special Investigation
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7981055; NCT06279221 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Japanese participants with alopecia areata: Japanese participants with alopecia areata
  Interventions: Drug: LITFULO

INTERVENTIONS:
Drug: LITFULO — as provided in real world practice

SUMMARY:
The objective of this Study is to confirm the safety during the long-term use of this drug and the effectiveness during the use of this drug under the actual use in the patients treated with this drug.

DETAILED DESCRIPTION:
This study is an open-label, multi-center, one arm prospective observational cohort study of patients receiving this drug. The investigators complete the CRF based on the information extracted from the medical record created in daily medical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

* Patients with alopecia areata who start receiving this drug for the first time after the contract date of this study
* Patients who have not participated in a clinical trial (clinical study) of this drug

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

* Patients previously enrolled in this study
* Patients with a history of treatment with this drug (including investigational product)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with alopecia areata who received LITFULO
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2030-06-25 (Estimated); Study Completion 2030-06-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with adverse events (AEs) | Baseline through year 3
Percentage of patients achieving SALT≤20 [SALT score (absolute value) 20 or less] | Baseline, evaluation at Week 12, Week 24 , Week 48, Week 78 , Week 104 , Week 130 , and Week 156 after the start of administration.
  The percentage of patients who achieved SALT ≤ 20 (absolute SALT score of ≤ 20) will be calculated at baseline (including the first day of treatment) and each evaluation time point after the start of treatment with this drug.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981055